CLINICAL TRIAL: NCT01535118
Title: National Allergies, Immunotherapy and RhinoConjunctivitis Survey in America
Brief Title: A Survey of Adults and Children With Allergic Rhinoconjunctivitis (MK-7243-021)
Acronym: AIRS
Status: Completed | Type: Observational
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: 7243-021
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Allergies; Immunotherapy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults and Children with Allergic Rhinoconjunctivitis (ARC): Adults and children with ARC who complete the survey

SUMMARY:
This study will gather information on allergic rhinoconjunctivitis from surveys completed by adults and children.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hay fever, rhinitis or nasal and/or eye allergies and display symptoms of sneezing, itching, watery eyes, nasal congestion, or other nasal or eye allergy symptoms over the past 12 months OR take any medication for their hay fever, rhinitis, nasal or eye allergies
* 5 years of age or older
* Have a telephone

Exclusion Criteria:

* If less than 18 years old and there is no adult available that is knowledgeable about the participant's health

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with ARC in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 2765 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

REFERENCES:
- [Result] Blaiss MS, Dykewicz MS, Skoner DP, Smith N, Leatherman B, Craig TJ, Bielory L, Walstein N, Allen-Ramey F. Diagnosis and treatment of nasal and ocular allergies: the Allergies, Immunotherapy, and RhinoconjunctivitiS (AIRS) surveys. Ann Allergy Asthma Immunol. 2014 Apr;112(4):322-8.e1. doi: 10.1016/j.anai.2014.02.006. PMID 24679733

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A national probablility sample of 2765 adults & children (age 5+) who had ever been diagnosed with hay fever, allergic rhinitis, rhinoconjunctivitis, nasal allergies or eye allergies & had nasal allergy symptoms in the past 12 months or had taken prescription medicine for allergies were interviewed by telephone about their condition & treatment.
Period: Overall Study
Arm/Group | Adults and Children With Allergic Rhinoconjunctivitis (ARC)
Started | 2765
Completed | 2765
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Adults and Children With ARC: Adults and children with ARC who complete the survey
Arm/Group | Adults and Children With ARC
Number analyzed (Participants) | 2765
Age, Customized [Number; unit: participants]
  5 to 11 years of age | 205
  12 to 17 years of age | 173
  18 to 24 years of age | 164
  25 to 34 years of age | 223
  35 to 44 years of age | 364
  45 to 54 years of age | 491
  55 to 64 years of age | 515
  65+ years of age | 597
  Don't Know/Refused | 33
Sex/Gender, Customized [Number; unit: participants]
  Female | 581
  Male | 333
  Unknown | 1851

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Daily Symptoms Due to Allergic Rhinoconjunctivitis (ARC)
Description: Participants were asked about the frequency and severity of ARC symptoms when allergies were at their worst. The percentages of participants who experienced different symptoms of ARC on a daily basis when allergies were at their worst were calculated.
Time Frame: Within 12 months prior to survey
Population: The analysis population consisted of all participants who responded to the survey.
Measure: Number; unit: percentage of participants
Arm/Group | Adults and Children With ARC
Number analyzed (Participants) | 2765
percentage of participants
  Nasal congestion or stuffed nose | 41
  Runny nose | 39
  Postnasal drip | 38
  Nasal itching | 29
  Red or itchy eyes | 26
  Facial pain or pressure | 12
  Throat itching | 17
  Repeated sneezing | 26

2. Primary Outcome: Percentage of Participants Who Experienced Work or School Absence Due to ARC in the Past 12 Months
Description: Participants were asked about the impact of ARC on loss of work and school time. The percentage of participants who experienced work or school absence due to ARC in the prior 12 months was calculated.
Time Frame: Within 12 months prior to survey
Population: The analysis population consisted of all participants who responded to the survey.
Measure: Number; unit: percentage of participants
Arm/Group | Adults and Children With ARC
Number analyzed (Participants) | 2765
percentage of participants | 35

3. Primary Outcome: Percentage of Participants Who Used Medication to Treat ARC in the Past 12 Months
Description: Participants were asked about prescription and over-the-counter medication use for ARC. The percentages of participants who used prescription and/or over-the-counter medication to treat ARC in the past 12 months were calculated.
Time Frame: Within 12 months prior to survey
Population: The analysis population consisted of all participants who responded to the survey.
Measure: Number; unit: percentage of participants
Arm/Group | Adults and Children With ARC
Number analyzed (Participants) | 2765
percentage of participants
  Prescription medications | 58
  Over-the-counter medications | 81

4. Primary Outcome: Percentage of Participants Who Received Immunotherapy to Treat ARC
Description: Participants who had ever received immunotherapy for ARC were asked about the type of immunotherapy - subcutaneous or sublingual - received. The percentage of participants who received immunotherapy to treat ARC was calculated.
Time Frame: Within 12 months prior to survey
Population: The analysis population consisted of all participants who responded to the survey.
Measure: Number; unit: percentage of participants
Arm/Group | Adults and Children With ARC
Number analyzed (Participants) | 2765
percentage of participants
  Subcutaneous allergy shots | 21
  Sublingual allergy drops | 2

5. Primary Outcome: Percentage of Participants Who Received Allergy Shots and Required Supplemental Prescription Allergy Medication
Description: Participants who received subcutaneous immunotherapy (allergy shots) were asked about prescription and over-the-counter medication use. The percentage of participants who received allergy shots to treat ARC, had not taken over-the-counter allergy medication and required supplemental prescription allergy medication for ARC was calculated.
Time Frame: Within 12 months prior to survey
Population: The analysis population consisted of all participants who responded to the survey, received immunotherapy (allergy shots) and had not taken over-the-counter allergy medication.
Measure: Number; unit: percentage of participants
Arm/Group | Adults and Children With ARC
Number analyzed (Participants) | 148
percentage of participants | 67

6. Secondary Outcome: Percentage of Participants Who Received Allergy Shots and Had a Co-morbid Condition of Asthma
Description: Participants were asked about co-morbid health conditions. The percentage of participants who had received allergy shots to treat ARC and had asthma was calculated.
Time Frame: Within 12 months prior to survey
Population: The analysis population consisted of all participants who responded to the survey and received allergy shots.
Measure: Number; unit: percentage of participants
Arm/Group | Adults and Children With ARC
Number analyzed (Participants) | 623
percentage of participants | 31

ADVERSE EVENTS:
Description: No formal reporting or recording of adverse events was conducted during this observational study.
Arm/Group | Adults and Children With ARC
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No